CLINICAL TRIAL: NCT01628718
Title: Adaptive Disclosure: A Combat-Specific PTSD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); University of Wyoming (Other); Boston University (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ariel Lang, PhD, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100322; W81XWH-10-1-0657 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2012-06-19; First posted 2012-06-27 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: OEF/OIF; Veterans; Psychotherapy; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent evaluator is blind to treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPT-C (Active Comparator): Cognitive Processing Therapy, cognitive version only (CPT-C) delivered in 12 60-minute one-on-one treatment sessions.
  Interventions: Behavioral: Cognitive Processing Therapy, cognitive version only (CPT-C)
- Adaptive Disclosure (AD) (Experimental): Adaptive Disclosure delivered in eight 90-minute one-on-one treatment sessions.
  Interventions: Behavioral: Adaptive Disclosure (AD)

INTERVENTIONS:
Behavioral: Adaptive Disclosure (AD) — Adaptive Disclosure (AD) is an eight-session fully manualized and piloted intervention designed specifically for Marines with PTSD stemming from a variety of traumatic deployment experiences. The approach combines imaginal exposure to activate trauma-related emotions and beliefs and cognitive and experiential techniques to modify maladaptive interpretations of the implication of various combat and operational experiences that contribute to symptoms and dysfunction.
  Other Names: AD
  Arms: Adaptive Disclosure (AD)
Behavioral: Cognitive Processing Therapy, cognitive version only (CPT-C) — Cognitive Processing Therapy (CPT) is a 12-session manualized therapy for posttraumatic stress disorder. The theory behind CPT conceptualizes PTSD as a disorder of "non-recovery" in which erroneous beliefs about the causes and consequences of traumatic events produce strong negative emotions and prevent accurate processing of the trauma memory and natural emotions emanating from the event. A significant contributor to the interruption of natural recovery process is the ongoing use of avoidance as a coping strategy. CPT incorporates trauma-specific cognitive techniques to help individuals with PTSD more accurately appraise these "stuck points" and progress toward recovery.
  Other Names: CPT-C
  Arms: CPT-C

SUMMARY:
The primary objective of this randomized controlled non-inferiority trial is to determine whether or not Adaptive Disclosure (AD), a new combat-specific psychotherapy for Post Traumatic Stress Disorder (PTSD), is as least as effective as Cognitive Processing Therapy, cognitive only version (CPT-C), in terms of its impact on deployment-related psychological health problems (specifically PTSD and depression) and functioning.

DETAILED DESCRIPTION:
Many Marines and Sailors return from deployment with mental health problems related to their experiences. One such problem is posttraumatic stress disorder (PTSD), which involves symptoms such as persistent unwanted memories of traumatic events, avoidance of reminders of the events, excessive watchfulness, jumpiness and irritability. Current therapies for PTSD focus chiefly on fear related to life-threat and were developed chiefly on civilians. We developed and piloted tested a psychological treatment for PTSD specifically for service members who suffer not only life-threat, but also traumatic loss and inner conflicts from morally challenging experiences. This intervention, Adaptive Disclosure (AD) is an eight-session PTSD treatment that helps Marines to identify unhelpful beliefs about a traumatic event and find ways to move forward. Preliminary clinical data suggests that AD is acceptable to Marines, feasible to implement, and safe and that it reduces PTSD and depression. The primary objective of this randomized controlled non-inferiority trial is to determine whether or not AD is as least as effective as Cognitive Processing Therapy, cognitive only version (CPT-C), which is an empirically validated and commonly used PTSD treatment.

We plan to recruit 266 Marines for this project. They will be randomly assigned to AD or CPT-C and followed during and after treatment. The groups will be compared on measures of mental health (particularly PTSD and depression), work-related functioning, trauma-related beliefs, coping and attitudes about mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current PTSD as diagnosed by the CAPS or subsyndromal PTSD (at least meeting criteria A and B) with distress and/or functional impairment as determined by the CAPS and review by study senior clinicians. Co-occurring disorders such as depression, anxiety, or treated substance abuse or dependence problems are permitted.
* Individuals expected to deploy two or more months from the time of referral and/or assessment are eligible. Anyone deploying sooner than that would be unable to complete the entire intervention and thus, are ineligible. Potential enrollees need not be presently deployable.
* Prospective enrollees must be willing to commit to 8 consecutive weekly sessions lasting up to 90 minutes in duration and to complete assessment materials.

Exclusion Criteria:

* Serious suicidality or homicidality that has required urgent or emergent evaluation or treatment within the past three months.
* A known, untreated substance abuse or dependence problem. Inclusion is possible if there is evidence that the individual has been afforded and is complying with treatment for the substance problem.
* Serious Axis I mental disorders (those that are normally incompatible with active military service), such as psychotic disorders or bipolar type I, are not eligible.
* Cognitive impairment that would interfere with one's ability to complete the intervention. If a potential participant performs below the mildly impaired range on WAIS-IV Digit Span or CVLT-2, the study neuropsychologist will review the case and make a clinical judgment based on review of testing and, in some cases, additional evaluation as to ability to participate.
* Concurrent enrollment in any cognitive-behavioral treatment, group therapy, or any other treatment that involves systematic disclosure of troubling deployment-related memories. Participants can continue current pharmacological treatment, marital counseling, or any supportive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-03; Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J Lang, PhD, Principal Investigator — Veterans Medical Research Foundation
Locations (2):
- United States (2):
  - Naval Hospital Camp Pendelton, Oceanside, California
  - Naval Medical Center San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litz BT, Rusowicz-Orazem L, Doros G, Grunthal B, Gray M, Nash W, Lang AJ. Adaptive disclosure, a combat-specific PTSD treatment, versus cognitive-processing therapy, in deployed marines and sailors: A randomized controlled non-inferiority trial. Psychiatry Res. 2021 Mar;297:113761. doi: 10.1016/j.psychres.2021.113761. Epub 2021 Jan 24. PMID 33540206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPT-C | Adaptive Disclosure (AD)
Started | 60 | 62
Completed | 33 | 37
Not Completed | 27 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPT-C | Adaptive Disclosure (AD) | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.29 (6.38) | 30.30 (6.43) | 29.80 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 54 | 56 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 36 | 41 | 77
  Other Race/Ethnicity | 24 | 21 | 45
Region of Enrollment [Number; unit: participants]
  United States | 60 | 62 | 122
PTSD severity as measured by the Clinician Administered PTSD Scale for DSM-IV (CAPS-IV) [Mean (Standard Deviation); unit: units on a scale] — CAPS Total Severity Score was calculated by summing frequency (0-4) and intensity (0-4) ratings for the 17 diagnostic symptoms. Total scores can be interpreted as follows: 0-19=asymptomatic/few symptoms, 20-39=mild PTSD/subthreshold, 40-59=moderate PTSD/threshold, 60-79=severe PTSD symptomatology, >80=extreme PTSD symptomatology. A 15-point change in CAPS total severity score has been proposed as a marker of clinically significant change.
  units on a scale | 76.53 (18.43) | 74.58 (19.25) | 75.54 (18.80)
PTSD severity as measures by the PTSD Checklist, military version (PCL-M) [Mean (Standard Deviation); unit: units on a scale] — A total score on the PCL-M is calculated by summing the 17 items (range 17-85), with higher scores indicating more severe symptoms.
  units on a scale | 62.47 (11.06) | 63.00 (11.45) | 62.74 (11.22)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status of Participants as Measured by the Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV)
Description: Proportion of patients recovered (meets Reliable Change Index (RCI) threshold and has change of at least 2SD from baseline to post-treatment), improved (meets positive RCI threshold), unchanged (does not meet RCI threshold) or deteriorated (meets negative RCI threshold) based on change in the CAPS-IV.
Time Frame: Pre-treatment (baseline), post-treatment (8-12 weeks)
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | CPT-C | Adaptive Disclosure (AD)
Number analyzed (Participants) | 60 | 62
Participants
  Recovered | 8 | 11
  Improved | 7 | 4
  Unchanged | 45 | 47
  Deteriorated | 0 | 0
Statistical Analysis 1: Comparison: CPT-C vs Adaptive Disclosure (AD); Null hypothesis: AD is inferior to CPT Alternative hypothesis: AD is non-inferior to CPT-C; Test type: Non-Inferiority — The NI margin for CAPS-IV scores was established a priori, based on a calculation of a reliable difference from baseline to posttreatment CAPS-IV scores from a previous trial (10 points). If the 95% confidence interval (CI) around the estimate does not contain the NI margin, we can reject the null hypothesis and accept the alternative hypothesis; p = .05, Regression, Linear — one-tailed; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-10.10 to 9.44] — Mean difference is the difference in mean CAPS-IV change scores (pre-post) between AD and CPT-C

ADVERSE EVENTS:
Time Frame: Period of study participation, which is time of enrollment through completion of the follow-up assessment, range approx. 36-40 weeks.
Arm/Group | CPT-C | Adaptive Disclosure (AD)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/62
Other Adverse Events (participants affected / at risk) | 4/60 | 10/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPT-C (N=60) | Adaptive Disclosure (AD) (N=62)
Alcohol poisoning (Psychiatric disorders) | 1 (1) | 0 (0)
Dissociative episode (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPT-C (N=60) | Adaptive Disclosure (AD) (N=62)
Increased psychiatric symptoms (Psychiatric disorders) | 1 (1) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Allergic reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT01628718/Prot_SAP_000.pdf